CLINICAL TRIAL: NCT06819007
Title: A Phase 3, Open-label, Multicenter, Randomized Trial of Trastuzumab Deruxtecan With Bevacizumab Versus Bevacizumab Monotherapy as First-line Maintenance Therapy in HER2-Expressing Ovarian Cancer (DESTINY-Ovarian01/ENGOT-ov89/GEICO144- O/GOG-3112/APGOT-OV13)
Brief Title: Study of Trastuzumab Deruxtecan With Bevacizumab Versus Bevacizumab Monotherapy for First-line Maintenance in HER2-Expressing Ovarian Cancer (DESTINY-Ovarian01)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-772; ENGOT-ov89 (Other Grant/Funding Number: ENGOT); GEICO144-O (Other Grant/Funding Number: ENGOT); GOG-3112 (Other Grant/Funding Number: GOG); APGOT-OV13 (Other Grant/Funding Number: APGOT)
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; epithelial ovarian cancer; HER2; Trastuzumab Deruxtecan; Bevacizumab
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — trastuzumab deruxtecan; Bevacizumab

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (Experimental): Participants will receive T-DXd in combination with bevacizumab
  Interventions: Drug: Trastuzumab Deruxtecan; Drug: Bevacizumab
- Treatment Arm B (Active Comparator): Participants will receive bevacizumab monotherapy
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — T-DXd will be administered at a dose of 5.4 mg/kg intravenously (IV) every 3 weeks (Q3W)
  Other Names: T-DXd; ENHERTU®
  Arms: Treatment Arm A
Drug: Bevacizumab — Bevacizumab will be administered at a dose of 15/mg/kg IV Q3W

SUMMARY:
This clinical trial is designed to evaluate the efficacy and safety of T-DXd in combination with bevacizumab versus bevacizumab monotherapy as first-line maintenance therapy, in participants with human epidermal growth factor 2 (HER2)-expressing (immunohistochemistry [IHC] 3+/2+/1+) advanced high-grade epithelial ovarian cancer.

DETAILED DESCRIPTION:
A non-randomized safety run-in phase will be conducted prior to randomization phase to assess the safety of T-DXd in combination with bevacizumab.

ELIGIBILITY:
Key Inclusion Criteria:

1. Sign and date the tissue prescreening informed consent form (ICF), prior to HER2 central testing. Sign and date the main ICF, prior to the start of any trial- specific qualification procedures. Consent to optional PGx prior to any PGx procedures. For participants in the safety run-in phase, a safety run-in ICF needs to be signed and dated prior to the start of any trial-specific qualification procedures.
2. Adults ≥18 years of age on the day of signing the ICF. Follow local regulatory requirements if the legal age of consent for trial participation is >18 years old.
3. Has histologically confirmed diagnosis of epithelial high-grade ovarian, fallopian tube or primary peritoneal carcinoma (including but not limiting to serous, endometrioid, clear cell, carcinosarcoma, mucinous).
4. Is newly diagnosed FIGO Stage III or IV.
5. Has HER2 expression per 2016 ASCO-CAP gastric cancer IHC scoring (3+/2+/1+) guidelines1 by prospective central testing. For participants in the safety run-in phase, HER2 expression assessed by either local (require using ASCO-CAP gastric cancer IHC scoring [IHC 3+/2+/1+] guidelines) or central assessment (if available) is acceptable. Submission of the pathology report is required for participants enrolled based on local HER2 IHC results.
6. Has adequate tumor tissue sample available for assessment of HER2 by central laboratory. Tumor tissue block or sufficient tissue slides are required for HER2 testing and retrospective HRD status determination. Participants in the safety run-in phase who are enrolled based on local HER2 IHC results are recommended to provide tumor tissue sample from the same specimen for central assessment.
7. Has a local HRD or breast cancer gene (BRCA) test result available. Participants with BRCA wildtype will have a local HRD test results, as applicable.
8. Has received standard of care bevacizumab in combination with front line platinum based chemotherapy as per approved indication and clinical guidelines and is eligible to continue single agent bevacizumab maintenance per standard of care and investigator discretion.

Key Exclusion Criteria:

1. Has ovarian, fallopian tube, or peritoneal cancer of non-epithelial origin.
2. Has a BRCA mutation as per local test.
3. Participant to receive PARP inhibitor as maintenance per standard of care and investigator discretion. Reasons for which the participant is not eligible for PARP inhibitor will be recorded in the eCRF as follows: HRD negative HRD positive with SD as best response after platinum HRD positive non-serous histology HRD tested, but inconclusive HRD positive but safety concern (safety concern to be specified).
4. Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug products and other monoclonal antibodies.
5. Previous Cerebral-Vascular Accident, Transient Ischemic Attack or Sub- Arachnoids Hemorrhage within 6 months prior to randomization.
6. Has evidence of bleeding diathesis or significant coagulopathy (in the absence of anticoagulation therapy).
7. Has a history of hemorrhagic disorders, abdominal fistula, gastrointestinal perforation, or active gastrointestinal bleeding within 6 months before randomization.
8. Evidence of active or ongoing bowel obstruction.
9. Has lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (eg, pulmonary emboli within 3 months of the trial randomization, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, pneumonectomy, etc.)
10. Has a history of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
11. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (ie pulmonary emboli within three months of the trial enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.), and any autoimmune, connective tissue or inflammatory disorders with potential pulmonary involvement (ie Rheumatoid arthritis, Sjogren's, sarcoidosis etc.), or prior pneumonectomy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 582 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival by Blinded Independent Central Review (BICR) in the HER2 IHC 3+/2+ population | From date of randomization to radiographic disease progression or death due to any cause, up to approximately 35 months
  Time from randomization to time of objective radiographic disease progression as assessed by BICR based on RECIST v1.1 or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival in the HER2 IHC 3+/2+ population | From date of randomization to death due to any cause, up to approximately 72 months
  Time interval from the date of randomization to the date of death due to any cause.
Progression Free Survival by BICR in the HER2 IHC 3+/2+/1+ population | From date of randomization to radiographic disease progression or death due to any cause, up to approximately 35 months
  Time from randomization to time of objective radiographic disease progression as assessed by BICR based on RECIST v1.1 or death due to any cause.
Overall Survival in the HER2 IHC 3+/2+/1+ population | From date of randomization to death due to any cause, up to approximately 72 months
  Time interval from the date of randomization to the date of death due to any cause.
Progression Free Survival by the investigator in HER2 IHC 3+/2+ population | From date of randomization to radiographic disease progression or death due to any cause, up to approximately 35 months
  Time from randomization to time of objective radiographic disease progression as assessed by the investigator based on RECIST v1.1 or death due to any cause.
Progression Free Survival by the investigator in HER2 IHC 3+/2+/1+ population | From date of randomization to radiographic disease progression or death due to any cause, up to approximately 35 months
  Time from randomization to time of objective radiographic disease progression as assessed by the investigator based on RECIST v1.1 or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (138):
- United States (20):
  - Scripps Clinic, La Jolla, California
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - Nancy N. & J.C Lewis Cancer & Research Pavillion- St. Josephs/ Candler Health System, Savannah, Georgia
  - Indiana University, Indianapolis, Indiana
  - Trials365 LLC, Shreveport, Louisiana
  - Greater Baltimore Medical Center, Towson, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Valley Health System, Paramus, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - UNC Hospital, Chapel Hill, North Carolina
  - Miami Valley Hospital South, Centerville, Ohio
  - Legacy Medical Group Gynecologic Oncology, Portland, Oregon
  - Providence Cancer Center Oncology, Portland, Oregon
  - St. Lukes University Health Network, Bethlehem, Pennsylvania
  - Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Avera Medical Group Gynecologic, Sioux Falls, South Dakota
- Genesiscare St Andrews Hospital, Adelaide, Australia
- Belgium (4):
  - UZ Leuven, Leuven
  - Groupe Sante CHC/Clinique du MontLegia, Liège
  - CHU UCL Namur, Namur
  - Cliniques Universitaires Saint-LUC, Woluwe-Saint-Lambert
- Brazil (9):
  - Oncocentro Belo Horizonte, Belo Horizonte
  - Centro De Pesquisas Clinica Reichow, Blumenau
  - Fundação Doutor Amaral Carvalho, Jaú
  - Liga Norte-Rio-Grandense Contra o Cancer, Natal
  - Centro Gaucho Integrado de Oncologia, Hematologia, Ensino e Pesquisa Hospital Mae de Deus, Porto Alegre
  - Irmandade Da Santa Casa De Misericordia De Porto Alegre, Porto Alegre
  - Ceon Pesquisas, Santo André
  - Fundacao Faculdade Regional De Medicina De Sao Jose Do Rio Preto, Sao Jose Rio
  - BP A Beneficencia Portuguesa de Sao Paulo, São Paulo
- Bulgaria (5):
  - Complex Oncology Center- Plovdiv EOOD, Plovdiv
  - MHAT Park Hospital EOOD, Plovdiv
  - MHAT Serdika EOOD, Sofia
  - UMHAT Sofiamed EOOD, Sofia
  - UMHAT Tsaritsa Yoanna ISUL EAD, Sofia
- China (26):
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Sichuan University West China Second University Hospital, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - The Second Hospital of Dalian Medical University, Dalian
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Harbin Medical University - Tumor Hospital, Haerbing
  - Hainan General Hospital, Haikou
  - Zhejiang Cancer Hospital, Hangzhou
  - Women's Hospital School of Medicine Zhejiang University, Hangzhoushi
  - Shandong Cancer Hospital, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Jiangxi Maternal and Child Health Hospital, Nanchang
  - Zhong Da Hospital, Southeast University, Nanjing
  - Guangxi Medical University Cancer Hopstial, Nanning
  - Fudan University Shanghai Cancer Center, Shanghai Shi
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Affiliated Hospital (Suzhou First People's Hospital), Suzhou
  - Shanxi Cancer Hospital, Taiyuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - Tongji Hospital Tongji Medical College of HUST, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
- Aarhus University Hospital, Aarhus, Denmark
- France (10):
  - Institut Bergonie, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Hopital Claude Huriez- CHU Lille, Lille
  - Centre Leon Berard, Lyon
  - CHU Montpellier, Saint Eloi, Montpellier
  - Hopital Prive Du Confluent, Nantes
  - Hopital Saint Joseph- Paris, Paris
  - Hospital Europeen Georges Pompidou, Paris
  - CRLCC Eugene Marquis, Rennes
  - CHU Saint Etienne, Saint-Etienne
- King George Hospital, Visakhapatnam, India
- Israel (5):
  - The Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (4):
  - Istituto Tumori Giovanni Paolo II Irccs Ospedale Oncologico Bari, Bari
  - Azienda Ospedaliera Per Lemergenza Cannizzaro, Catania
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Istituto Nazionale Tumori Regina Elena Irccs, Roma
- Japan (16):
  - Hyogo Cancer Center, Akashi
  - National Cancer Center Hospital, Chūōku
  - Fukushima Medical University Hospital, Fukushima
  - Saitama Medical University International Medical Center, Hidaka-Shi
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Kurume University Hospital, Kurume-shi
  - Aichi Cancer Center Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hosptial, Okayama
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Osakasayama-shi
  - NHO Hokkaido Cancer Center, Sapporo
  - Iwate Medical University Hospital, Shiwa-Gun
  - Shizuoka Cancer Center, Sunto-gun
  - Mie University Hospital, Tsu
  - Yamagata University Hospital, Yamagata
- Malaysia (4):
  - Hospital Sultan, Johor Bahru
  - Sarawak General Hospital, Kuching
  - HOSPITAL KUALA LUMPUR(HKL) Kuala, Lumpur
  - National Cancer Institute / Institut Kanser Negara, Putrajaya
- Mazowiecki Szpital Wojewodzki W Siedlcach SP Zoo, Siedlce, Poland
- Romania (4):
  - Gral Medical S.R.L, Bucharest
  - Medeuropa SRL, Bucharest
  - Memorial Healthcare International SRL, Bucharest
  - Medeuropa SRL, Oradea
- National University Hospital, Singapore, Singapore
- South Korea (10):
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Goyang-si
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary'S Hospital, Seoul
- Spain (7):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Clinica Universidad de Navarra (MAD), Pamplona
  - Clinica Universidad de Navarra (Calle Marquesado de Santa Marta), San Blas-Canillejas
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (7):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Linkou Taoyuan
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - MacKay Memorial Hospital- Taipei Branch, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/